CLINICAL TRIAL: NCT00234377
Title: A 12-week International, Multicenter, Open Label, Non-comparative Study to Evaluate the Feasibility of Switching Any Antipsychotic Treatment to Sustained-release Quetiapine Fumarate (SEROQUEL®) in Patients With Schizophrenia
Brief Title: Seroquel Switching Study: Feasibility of Switching Any Antipsychotic Treatment to Seroquel in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1444C00147
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Seroquel SR

SUMMARY:
The purpose of this study is to document the clinical benefit of quetiapine (Seroquel) sustained release (SR) after switching from another ongoing antipsychotic treatment, regardless of the reason for the switch.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Patients who in their own and/or in the Investigator's opinion, consider ongoing antipsychotic treatment inadequate, because of insufficient efficacy and/or tolerability.
* Female patients of childbearing potential must have a negative serum pregnancy test at enrolment and be willing to use a reliable method of birth control, ie, barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device, or tubal ligation during the study.
* Able to understand and comply with the requirements of the study, as judged by the Investigator.

Exclusion Criteria:

* Meeting the criteria for any other (than schizophrenia) Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) Axis I diagnosis, concomitant organic mental disorder or mental retardation.
* Substance abuse or dependence as defined by DSM-IV and not in full remission. A urine drug screen test will be performed. The Investigator will evaluate the results along with medical history to determine if the patient meets DSM-IV criteria for substance abuse or dependence.
* Risk of transmitting human immunodeficiency virus (HIV) or hepatitis B, via blood or other body fluids, as judged by the Investigator.
* Patients who, in the opinion of the Investigator, pose an imminent risk of suicide or a danger to self or others.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550
Dates: Start 2004-11; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who have an improved clinical benefit based on assessment of clinical efficacy in combination with assessment of tolerability

SECONDARY OUTCOMES:
The change from baseline in Clinical Global Impression (CGI)-CB score
Change from baseline in Positive and Negative Syndrome Scale (PANSS) total score

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca CNS Medical Science Director, MD, Study Director — AstraZeneca
Locations (27):
- Canada (10):
  - Research Site, Vancouver, British Columbia
  - Research Site, Aurora, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Orléans, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Saint-Laurent, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Prince Albert, Saskatchewan
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Mikkeli
  - Research Site, Turku
- Germany (10):
  - Research Site, München, Bavaria
  - Research Site, Göttingen, Lower Saxony
  - Research Site, Aachen, North Rhine-Westphalia
  - Research Site, Saarbrücken, Saarland
  - Research Site, Aachen
  - Research Site, Göttingen
  - Research Site, Halle
  - Research Site, Homburg
  - Research Site, Jena
  - Research Site, München
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyula
  - Research Site, Székesfehérvár

REFERENCES:
- [Derived] Ganesan S, Agambaram V, Randeree F, Eggens I, Huizar K, Meulien D; Study 147 Investigators. Switching from other antipsychotics to once-daily extended release quetiapine fumarate in patients with schizophrenia. Curr Med Res Opin. 2008 Jan;24(1):21-32. doi: 10.1185/030079908x253384. PMID 18021496